CLINICAL TRIAL: NCT02659722
Title: A Multi-Center Prospective Study of Vertebral Technologies, Inc. (VTI) InterFuse® S and InterFuse® T for the Treatment of Scoliosis, Spondylolisthesis and Degenerative Disc Disease.
Brief Title: InterFuse® S and T for the Treatment of Scoliosis, Spondylolisthesis and Degenerative Disc Disease (DDD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vertebral Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VTI-012
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Scoliosis; Back Pain
Keywords: INTERVERTEBRAL DISC DEGENERATION; Bone Disease; Musculoskeletal disease; Spinal disease
MeSH Terms: conditions — Scoliosis; Back Pain; Intervertebral Disc Degeneration; Bone Diseases; Musculoskeletal Diseases; Spinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: InterFuse — TRansforaminal or Posterior placement of an InterFuse S and/or T device, in combination with approved posterior fixation
  Other Names: InterFuse S; InterFuse T; Modular Lumbar Interbody Fusion; Expandable cage

SUMMARY:
The primary objective of this prospective, post-market study is to collect data to assess the long term outcome of a broad contact modular interbody device in the form of the InterFuse S™ or InterFuse T™ device in patients undergoing long construct fusion for degenerative disc disease and/or scoliosis. Comparisons will be made with published historical data..

DETAILED DESCRIPTION:
The primary objective of this prospective, post-market study is to collect data to assess the long term outcome of a broad contact modular interbody device in the form of the InterFuse S™ or InterFuse T™ device in patients undergoing long construct fusion for degenerative disc disease and/or scoliosis. While there is no concurrent control population, there is ample historical control data to be used for comparison.

The study will include up to two hundred (200) patients, up to 10 centers, and provide a prospective evaluation of the InterFuse "T" and/or InterFuse "S" Interbody Fusion System. Primary endpoints will be assessed at twelve months post-surgery. All patients enrolled in the study will be followed for at least 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patients has a planned fusion construct of at least five levels and will have the InterFuse (S) or (T) planned for L5-S1 and/or L4-L5.

  2. The patient has documented conservative (non-operative) treatment for at least 6 months.

  3. The patient has a VAS score of ≥ 60 mm for Back and/or Leg. 4. The patient has an ODI ≥ 40%. 5. The general condition of the patient is appropriate for surgery, as evaluated by the Investigator.

  6. The patient is willing and able to comply with study requirements. 7. The patient has agreed to participate in the study

Exclusion Criteria:

* 1. The patient has undergone any prior spinal fusion surgery at the proposed treatment level(s). Previous non-fusion surgery at the proposed treatment level(s) is acceptable.

  2. The patient has osteoporosis or severe osteopenia as determined by the Investigator. A clinical SCORE calculator may be utilized for females over 40 years of age.

  3. The patient has grade 2 or higher spondylolisthesis or retrolisthesis at the affected level(s).

  4. The patient has known neoplastic disease other than skin cancer. 5. The patient has a Body Mass Index (BMI) of greater than 40; BMI = wt (kg)/ht2 (m2).

  6. The patient has an active infection. 7. The patient is pregnant or is planning on becoming pregnant in the next two years.

  8. The patient is mentally ill or has a history of drug abuse or severe depression/ psychosocial issues.

  9. The patient has a known allergy to polyether ether ketone (PEEK), stainless steel or tantalum.

  10. The patient is currently enrolled in an investigational spine study. 11. The patient has rheumatoid arthritis, ankylosing spondylitis or other autoimmune disease.

  12. The patient has symptomatic fibrous arachroiditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The protocol includes skeletally mature patients both male and female, 18 to 89 years old, with degenerative disc disease (DDD) and/or scoliosis and a planned fusion of at least five levels.. DDD is defined as discogenic back pain with degeneration of the disc confirmed by patient history and radiographic studies.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-06 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
disc height retention | 24 months
  loss of restored disc height over time
Complications | 24 months
  Migration, subsidence, hardware lossening and others
Lordosis | 24 months
  retention of restored degree of lordosis
Fusion | 24 months
  Speed of fusion

SECONDARY OUTCOMES:
Pain and function Scores | 24 months
  Visual Analog Scale (VAS) leg and back (at rest and active)
Scoliosis Research Society (SRS) Scores | 24 months
  Scoliosis Research Society Scores
Complications II | 24 months
  re-admission rate and re-operation rate

CONTACTS AND LOCATIONS:
Overall Officials: William Lavelle, MD, Principal Investigator — SUNY Unpstate
Locations (1):
- SUNY Upstate, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Presentations by investigator(s) at scientific meetings, submission of manuscript to peer reviewed journal